CLINICAL TRIAL: NCT03180723
Title: Effect of Rituximab in Treatment of Primary Membranoproliferative Glomerulonephritis
Brief Title: Effect of Rituximab in Treatment of Membranoproliferative Glomerulonephritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Hassan Farghally, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMPGN
Record Dates: First submitted 2017-06-03; First posted 2017-06-08 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Membranoproliferative Glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative | interventions — Rituximab; Cyclosporine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Rituximab is given in 2 doses (1 gm each dose) to a group of15 patients with primary membranoproliferative glomerulonephritis at (0 - after 2 weeks)
  Interventions: Drug: Rituximab
- control group (Active Comparator): Cyclosporine is given orally in a dose of 2mg/kg/d for 3 months to another group of patients with primary membranoproliferative glomerulonephritis.
  Interventions: Drug: Cyclosporin

INTERVENTIONS:
Drug: Rituximab — Intravenous injection
  Arms: study group
Drug: Cyclosporin — Oral tablets
  Arms: control group

SUMMARY:
Type I membranoproliferative glomerulonephritis (MPGN) is a relatively uncommon glomerular disease, constituting 1.8% of renal biopsies performed in Rochester, minnesota, United States of America, at the Mayo Clinic, between 1993 and 2008. The prognosis of idiopathic Type I MPGN is relatively poor. Recently, Irish series, slightly more than 50% of patients developed end stage renal disease after a mean follow up of 14 years . The disease may recur after renal transplantation . High-dose glucocorticoids have been used to treat this disease in children but there is no established treatment in adults.

DETAILED DESCRIPTION:
Type I MPGN is associated with a variety of disorders, including hepatitis, especially hepatitis C, cryoglobulinemia, monoclonal gammopathies, systemic lupus erythematosus, and bacterial endocarditis or other chronic bacterial infections . Idiopathic Type I MPGN is rare. Biopsy samples usually stain for C3 and properdin. However, immunoglobulin G is also present in most cases, especially if the biopsy is performed early in the course of the disease suggesting antibody production as a possible therapeutic target.

Rituximab is a chimeric murine/human immunoglobulin g1 kappa monoclonal antibody targeting the cluster of differentiation 20 antigen found on pre-B and mature B lymphocytes, but not on hematopoietic stem cells, pro-B cells, normal plasma cells or the cells of other normal tissues. In the United States it was approved by the US Food and Drug Administration in 1997 for non-Hodgkin's lymphoma and was later approved for rheumatoid arthritis. Intravenous administration of rituximab results in rapid, selective, prolonged B cell depletion.

Anecdotal reports have demonstrated the efficacy of rituximab in treating MPGN secondary to chronic lymphocytic leukemia. Rituximab has also been shown to be effective in patients with MPGN related to a monoclonal gammopathy.

In an open label trial with rituximab, six patients with MPGN type I were treated with rituximab 1000 mg on days 1 and 15 and followed for 1 year. Proteinuria fell in all patients, at all time points, after rituximab administration. Renal function did not change.

ELIGIBILITY:
Inclusion Criteria:

1. MPGN either native/renal transplant kidneys with biopsy last 3 years.
2. Age > 18 years.
3. Urinary protein to creatinine ratio > 1.0 in a 24-hour urine collection, despite angiotensin converting enzyme inhibitor/angiotensin receptor blocker treatment.
4. Patients need to be treated with an ACEI and/or ARB, for at least 3 months prior to enrollment with the systolic blood pressure < 140 mm Hg for at least 75% of readings.
5. Women must be post-menopausal, surgically sterile or practicing a medically approved method of contraception.
6. Patients intolerant of ACE inhibitors/ARBs may enter the study without being treated with these agents.
7. Estimated glomerular filtration rate ≥ 25 ml/min per 1.73m^2 in the presence of ACE inhibitor/ARB therapy. The GFR will be estimated using the 4 variable Modification of Diet in Renal Disease (MDRD) equation/National Kidney Foundation - Chronic Kidney Disease (NKF-CKD) guidelines.
8. Adequate liver function.
9. Negative serum pregnancy test (for women of child bearing age).

Exclusion Criteria:

1. Age <18 years.
2. Secondary MPGN.
3. Presence or suspicion of active infection.
4. Pregnancy.
5. Concomitant malignancies, Major psychiatric disorder. Significant cardiac or pulmonary disease and any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory suspicion of a disease/condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
6. Laboratory Exclusion Criteria (Screening):

   * Hemoglobin:< 8.5 gm/dL
   * Platelets:< 100,000/mm
   * Total bilirubin, Aspartate amino transferase, alkaline phosphatase > 2.5 x Upper Limit of Normal unless related to primary disease
   * Positive Hepatitis B or C serology
   * Positive human immunodeficiency virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
effect of Rituximab on proteinuria | 3 months
  measured through urinary protein/ creatinine ratio

REFERENCES:
- [Background] Dillon JJ, Hladunewich M, Haley WE, Reich HN, Cattran DC, Fervenza FC. Rituximab therapy for Type I membranoproliferative glomerulonephritis. Clin Nephrol. 2012 Apr;77(4):290-5. doi: 10.5414/cn107299. PMID 22445472